CLINICAL TRIAL: NCT04839848
Title: Mesh and Fixation Combinations in the Lichtenstein Groin Hernioplasty: Association With Chronic Postoperative Pain. A Swedish Hernia Registry Study.
Brief Title: Chronic Postoperative Pain After the Lichtenstein Groin Hernioplasty
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other); Swedish Hernia Registry (Unknown)
Responsible Party: Principal Investigator, Bengt Novik, MD, SSOD, Karolinska Institutet
Other Study IDs: Bengan V
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Hernia, Inguinal; Hernia, Femoral; Postoperative Pain; Chronic Pain; PROM; Suture Related Complication
Keywords: Swedish Hernia Registry; Lichtenstein; Surgical mesh; Surgical sutures
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Femoral; Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (5):
- Permanent suture: Mesh fixation with permanent suture
  Interventions: Device: Lichtenstein mesh repair
- Long-term absorbable: Mesh fixation with long-term absorbable suture
  Interventions: Device: Lichtenstein mesh repair
- Short-term absorbable: Mesh fixation with short-term absorbable suture
  Interventions: Device: Lichtenstein mesh repair
- Fibrin glue: Biologic glue/sealant produced from human donor blood
  Interventions: Device: Lichtenstein mesh repair
- Progrip: Pre-fabricated absorbable fixation hooks, integrated in mesh. Progrip is a registered trademark owned by Medtronic
  Interventions: Device: Lichtenstein mesh repair

INTERVENTIONS:
Device: Lichtenstein mesh repair — A groin hernia repair, reinforced by synthetic mesh. The mesh is affixed with sutures

SUMMARY:
The study attempts to quantify the relative risks for chronic postoperative inguinal pain (CPIP) after Lichtenstein repair of groin hernia, depending on mesh type and fixation suture material.

For this purpose the investigators will analyze data from the Swedish Hernia Registry (SHR).

DETAILED DESCRIPTION:
This is an open cohort study design where the investigators will analyze existing data that have been prospectively collected in SHR, which covers > 95% of all groin hernia repairs in Sweden. The large database enables assessment of the relative risks for CPIP depending on in particular mesh and mesh fixation, adjusted for other plausible risk factors.

Each participant was entered at the date of surgery, when demographic and intraoperative data were registered. One year postop, each patient was sent a questionnaire focusing on present pain.

ELIGIBILITY:
Inclusion Criteria:

All Lichtenstein and similar open mesh repairs that have been registered in the SHR from September 1, 2012, until December 31, 2018.

Exclusion Criteria:

* Laparoscopic repairs.
* Preperitoneal open repairs.
* Pure suture repairs
* Patients not having a 10-digit state-assigned Patient Identification Number.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An unselected, consecutive nationwide cohort during 7 years, with a 1-year follow-up
Sampling Method: Non-Probability Sample
Enrollment: 80733 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
CPIP | 1 year
  Chronic postoperative inguinal pain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Novik B, Nordin P, Skullman S, Dalenback J, Enochsson L. More recurrences after hernia mesh fixation with short-term absorbable sutures: A registry study of 82 015 Lichtenstein repairs. Arch Surg. 2011 Jan;146(1):12-7. doi: 10.1001/archsurg.2010.302. PMID 21242440
- [Background] Novik B, Hagedorn S, Mork UB, Dahlin K, Skullman S, Dalenback J. Fibrin glue for securing the mesh in laparoscopic totally extraperitoneal inguinal hernia repair: a study with a 40-month prospective follow-up period. Surg Endosc. 2006 Mar;20(3):462-7. doi: 10.1007/s00464-005-0391-3. Epub 2006 Jan 19. PMID 16424986
- [Background] Franneby U, Gunnarsson U, Andersson M, Heuman R, Nordin P, Nyren O, Sandblom G. Validation of an Inguinal Pain Questionnaire for assessment of chronic pain after groin hernia repair. Br J Surg. 2008 Apr;95(4):488-93. doi: 10.1002/bjs.6014. PMID 18161900
- [Background] Olsson A, Sandblom G, Franneby U, Sonden A, Gunnarsson U, Dahlstrand U. The Short-Form Inguinal Pain Questionnaire (sf-IPQ): An Instrument for Rating Groin Pain After Inguinal Hernia Surgery in Daily Clinical Practice. World J Surg. 2019 Mar;43(3):806-811. doi: 10.1007/s00268-018-4863-8. PMID 30478683
- [Background] Novik B, Sandblom G, Ansorge C, Thorell A. Association of Mesh and Fixation Options with Reoperation Risk after Laparoscopic Groin Hernia Surgery: A Swedish Hernia Registry Study of 25,190 Totally Extraperitoneal and Transabdominal Preperitoneal Repairs. J Am Coll Surg. 2022 Mar 1;234(3):311-325. doi: 10.1097/XCS.0000000000000060. PMID 35213495